CLINICAL TRIAL: NCT02360358
Title: A Phase II Randomized Multicenter Study on Efficacy and Safety of Cultured Autologous Skin (Tiscover®) and Acellular Dermal Matrix (AS210) in Chronic (Arterio-)Venous Ulcers
Brief Title: Autologous Skin Substitute for Chronic Leg/Foot Ulcers.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow inclusion
Sponsor: Chantal Blok (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Chantal Blok, trial coordinator, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIS2012
Record Dates: First submitted 2015-01-29; First posted 2015-02-10 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Varicose Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- autologous cultured skin (Experimental): autologous cultured skin patches (Tiscover) is applied on wound in 2-step procedure with 1 week interval. Dosage: number of patches depends on wound size. Application week 0 is removed after one week (week1). Week 1: wound is completely covered with new Tiscover patches.
  Interventions: Drug: Tiscover
- acellular donor dermis (Active Comparator): acellular donor dermis (AS210) is applied on wound in 2-step procedure with 1 week interval. Dosage: number of patches depends on wound size.
  Application week 0 is removed after one week (week1). Week 1: wound is completely covered with new AS210 patches.
  Interventions: Other: AS210

INTERVENTIONS:
Drug: Tiscover — two step procedure, week 0 and week1. Dosage depends on wound size.
  Other Names: autologous skin substitute
  Arms: autologous cultured skin
Other: AS210 — two step procedure, week 0 and week1. Dosage depends on wound size.
  Other Names: Acellular donor dermis
  Arms: acellular donor dermis

SUMMARY:
A prospective, multicenter, randomised controlled phase II study in which patients with therapy resistant (arterio-) venous leg/foot ulcers are treated with Tiscover® (test group) or with AS210 (control group) to determine the safety and relative efficacy of both products.

DETAILED DESCRIPTION:
Multicenter, randomised clinical trial in out patient in which patients with chronic (arterio-) venous leg/foot ulcers are treated with an autologous cultured human living skin substitute (Tiscover®: test group) or with Acellular donor dermis (AS210: control group). During a pre-inclusion evaluation period of 4 weeks (non healing) chronicity of ulcer is ensured (ulcer size change of < 30%). To determine ulcer type ABI, Doppler and CEAP is performed.

The test group will receive 2 applications of Tiscover®. Week 0: wound activating pre-treatment, application of at least one quarter of the wound surface. Week 1: removal of patches, application of patches on total wound surface.

The control group (16 patients) will follow the same application protocol.

ELIGIBILITY:
Inclusion criteria:

* Have a (arterio) venous leg ulcer (VLU) between the knee and ankle (at or above the malleolus), or on foot (not plantar side of the foot) with a surface area ≥ 1.0 cm2 and ≤ 40.0 cm2
* Venous insufficiency confirmed by duplex Doppler ultrasound examination for valvular or venous incompetence.
* Arterial supply adequacy confirmed (ABPI ≥ 0.6 and ≤ 1.3)
* Target ulcer involves a full thickness skin loss, but WITHOUT exposure of tendon, muscle, or bone. Ulcer depth < 1 cm
* Target ulcer duration ≥ 12 weeks but ≤ 15 years
* Acceptable state of health and nutrition
* Mobile, at least able to walk with medical walker, and able to return for required treatments and study evaluations

Exclusion Criteria:

* History of anaphylaxis, serum sickness, or erythema multiforme reaction to bovine serum proteins, gentamycin.
* Therapy with another investigational agent within thirty (30) days of Screening, or during the study.
* A target ulcer of non-venous etiologies (e.g., sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma gangrenosum, vasculopathic or vasculitic).
* Documented history of osteomyelitis at the target wound location within 6 months preceding the Screening Visit.
* Refusal of or inability to tolerate compression therapy.
* Therapy of the target ulcer with autologous skin graft, Apligraf™, or Dermagraft™ within 30 days preceding the Screening Visit.
* History of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancers).
* >30% change of wound size in 4 weeks or confirmed by historical data
* Presence of deep vein thrombosis or contra indication for compression therapy
* Severe co-morbidity reducing life expectance to < 1 year
* Use of oral corticosteroids and/or cytostatics >20 mg/per day;
* Severe infection of ulcer, active cellulitis, osteomyelitis
* Severe malnutrition
* Uncontrolled diabetes mellitus, HbA1c > 12% (108 mmol/mol)
* Anaemia Hb <6 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with complete wound closure after 26 weeks. | 26 weeks
  The primary objective of this study is to demonstrate the superiority of Tiscover® compared to AS210 for achieving wound healing in subjects with a chronic (arterio) venous leg or foot ulcer.

SECONDARY OUTCOMES:
Time in days to complete wound closure from baseline. | 12 weeks
• Proportion of subjects with complete wound closure at each of the 12 treatment weeks. | 12 weeks
Percentage of wound closure | 12 and 26 weeks
Proportion of subjects with durable wound healing over the 3 months following complete wound closure | 3 months and 6 months follow up
Wound size reduction | 12 and 26 weeks
  The percentage of reduction in wound area
Pain | week 0, 1,2,4,8,12, 26 weeks and follow up
  Measured with VAS Pain scale
Quality of Life | Week 0, 12, 26 weeks and follow up
  Measured with SF 36
Number of SAE | 12, 26 weeks and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gibss, Prof.dr., Study Chair — VU medical center, department of dermatology
Locations (5):
- Netherlands (5):
  - Centrum Oosterwal, Alkmaar
  - Flevo Ziekenhuis, afdeling dermatologie, Almere Stad
  - VU University Medical center, Amsterdam
  - St. Fransiscus Gasthuis, Rotterdam
  - Isala Ziekenhuis, dermatologie, Zwolle